CLINICAL TRIAL: NCT05428982
Title: The Effect of Postoperative Modified Trendelenburg Position to Decrease Shoulder Pain After Laparoscopic Hysterectomy: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 65055
Record Dates: First submitted 2022-06-07; First posted 2022-06-23 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-07

CONDITIONS: Post Operative Pain; Shoulder Pain; Gynecologic Disease
Keywords: Modified Trendelenburg, Shoulder Pain, Laparoscopic hysterectomy
MeSH Terms: conditions — Pain, Postoperative; Shoulder Pain; Genital Diseases, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postoperative Modified Trendelenburg group (Experimental): Patients underwent the laparoscopic hysterectomy were positioned in a Modified Trendelenburg position (20 °) postoperative for 6 hours
  Interventions: Procedure: Postoperative Modified Trendelenburg position
- Control (No Intervention): Patients underwent the laparoscopic hysterectomy were positioned in a neutral position

INTERVENTIONS:
Procedure: Postoperative Modified Trendelenburg position — Patients underwent the laparoscopic hysterectomy were positioned in a Modified Trendelenburg position (20 °) postoperative for 6 hours at ward.
  Arms: Postoperative Modified Trendelenburg group

SUMMARY:
Laparoscopic surgery is commonly used procedure in diagnostic and treatment including Hysterectomy. Post laparoscopic shoulder pain is common side effect mostly occur after surgery. Postoperative Trendelenburg position might decrease pain by reducing the mechanical pressure of CO2 on the diaphragm. Maintaining the patient in Trendelenburg for 6 hours postoperatively will decrease postoperative shoulder pain.

DETAILED DESCRIPTION:
After laparoscopic hysterectomy surgery, Patients in intervention group were positioned in a Modified Trendelenburg position (20 °) postoperative for 6 hours because of the limitation of this study cannot positioned in Trendelenburg position.

A modified Trendelenburg position is head and trunk of patient were in neutral position while hips and lower extrimities were raised at 20 degree.

In control group were in neutral position. All patients were asked shoulder pain score at ward, 6 , 12, 24 hours after postoperative Modified Trendelenburg position for 6 hours

ELIGIBILITY:
Inclusion Criteria:

* Female patient age between 30-65 years
* American Society of Anesthesiologist (ASA) physical status I or II
* Scheduled for operative laparoscopic hysterectomy with abdominal incisions measuring less than 1 cm in size
* Can speak and understand Thai language

Exclusion Criteria:

* Pregnant women
* Conversion procedure to open abdominal surgery
* Patients with postoperative abdominal drainage
* Surgery duration more than 3 hours
* Gynecologic malignancy surgery
* Patients with history of chronic shoulder pain
* Patients with history of previous shoulder surgery
* Inability to accurately express pain
* Patients with history of Gastroesophageal reflux disease or chronic gastritis
* Patients with history of cardiovascular or pulmonary disease
* Patients with history of venous thrombosis
* Morbid obesity BMI > 40 kg/m2
* Patients with history of increase intracranial pressure
* Patients with history of increase intraocular pressure
* Patients with liver and/or kidney disease
* NSAIDs and/or Paracetamol and/or Morphine allergy
* Current corticosteroid use
* Patients who use current analgesic drugs and don't want to quit while stay in the hospital
* Psychiatric disorder
* Intellectual disorder
* Postoperative length in hospital less than 24 hours

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Comparison of shoulder pain score | at ward, 6 , 12, 24 hours after postoperative Modified Trendelenburg position for 6 hours
  Comparison of shoulder pain score at 6 hours after postoperative Modified Trendelenburg position for 6 hours Using Numerical rating scale 0-10, 0 mean no pain, 10 mean worst pain

SECONDARY OUTCOMES:
Comparison of nausea vomiting score | at ward, 6 , 12, 24 hours after postoperative Modified Trendelenburg position for 6 hours
  Comparison of nausea vomiting score at ward, 6 , 12, 24 hours after postoperative Modified Trendelenburg position for 6 hours Nausea vomiting score grading : 1. None mean no symptom, 2. Mild mean only nausea, not required antiemetic drugs 3.Moderate mean have symptom of nausea and vomiting and required antiemetic drugs 4.Severe mean have symptom of nausea and vomiting and required antiemetic drugs more than 1 time
Total amount of antiemetic drugs in 24 hours postoperatively | 24 hours postoperatively
  Total amount of antiemetic drugs in 24 hours postoperatively
Comparison of upper abdominal pain score | at ward, 6 , 12, 24 hours after postoperative Modified Trendelenburg position for 6 hours
  Comparison of upper abdominal pain score at ward, 6 , 12, 24 hours after postoperative Modified Trendelenburg position for 6 hours Using Numerical rating scale 0-10, 0 mean no pain, 10 mean worst pain
Comparison of lower abdominal pain score | at ward, 6 , 12, 24 hours after postoperative Modified Trendelenburg position for 6 hours
  Comparison of lower abdominal pain score at ward, 6 , 12, 24 hours after postoperative Modified Trendelenburg position for 6 hours Using Numerical rating scale 0-10, 0 mean no pain, 10 mean worst pain

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand